CLINICAL TRIAL: NCT04637750
Title: Evaluation of the Effectiveness of a Low-cost Informative Intervention to Improve the Appropriate Prescription of Proton Pump Inhibitors in Older People in Primary Care: a Cluster- Randomized Controlled Study
Brief Title: Proton Pump Inhibitors (PPI): a Study to Improve Appropriate Prescriptions in the Elderly
Acronym: LAPTOP-PPI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mario Negri Institute for Pharmacological Research (Other)
Collaborators: IRCCS Multimedica (Other); Federico II University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GR-2016-02361198
Record Dates: First submitted 2020-11-09; First posted 2020-11-20 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2021-09

CONDITIONS: Proton Pump Inhibitor; Primary Care
Keywords: Proton pump inhibitors; prescription appropriateness
MeSH Terms: interventions — Early Intervention, Educational

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Educational intervention (Experimental): Randomised GPs will receive the low cost informative intervention composed by a practitioner-focused letter plus leaflet for patients
  Interventions: Behavioral: Educational intervention
- Control group (No Intervention): GPs not receiving any informative intervention

INTERVENTIONS:
Behavioral: Educational intervention — The GPs randomized to the intervention arm will receive a feedback informing on their absolute number of patients treated with at least one PPI during the baseline period and if they have been prescribed above or below the median of appropriate prescriptions rate in their local area. They will be also provided with a scientific document including technical details on AIFA reimbursement criteria (NOTA 1 and 48), short hints about adverse events related to PPI long- term use in older patients and recommendation on how to discontinue PPI therapy (i.e. gradual step down administration to avoid paradoxical effect).
  Arms: Educational intervention

SUMMARY:
Proton Pump Inhibitors(PPIs) are the leading evidence-based therapy for upper gastrointestinal disorders and prevention of antiplatelet or non-steroidal anti-inflammatory drugs induced ulcer. In Italy in 2015 nearly 3,5 millions of people were treated with PPI. Despite the extensive literature regarding PPI adverse event, their inappropriate prescription rate is still increasing, and Campania and Lombardy region are at the highest level. For this reason a cluster-randomised controlled trial will be performed, in order to evaluate if a low-cost informative intervention addressed to GPs is effective in improving PPIs prescription in older people. The threshold will be defined according to the distribution of the rate of appropriate PPI prescriptions for a 6 months lag time starting 1 year before randomisation (baseline assessment).

DETAILED DESCRIPTION:
A cluster-randomized controlled trial will be performed in order to evaluate if a low-cost informative intervention addressed to GPs is effective in improving PPIs prescription in older people. All GPs of the Local Health Unit (LHU) of Caserta (southern Italy) and Bergamo (northern Italy) will be invited to participate to the study, because Caserta and Bergamo represent the areas with the highest level of inappropriate PPI prescription rate. All GPs involved in the study will receive an invitation letter illustrating the study purpose and containing information about aggregated data on PPI prescriptions out of AIFA reimbursement criteria in Italy and their local area. The GPs randomized to the intervention arm will also receive a feedback informing on their absolute number of patients treated with at least one PPI during the baseline period and if they have been prescribed above or below the median of appropriate prescriptions rate in their local area. They will be also provided with a scientific document including technical details on AIFA reimbursement criteria (NOTA 1 and 48), short hints about adverse events related to PPI long- term use in older patients and recommendation on how to discontinue PPI. After 4 months GPs will also receive a patient-focused intervention leaflet and poster for patients about their medicines: what are the PPI and their possible side effects, nutritional and behavioral advices to prevent gastric and reflux problems and how to step down the treatment. The appropriateness of PPI prescriptions will be defined according to the Italian Medicines Agency (AIFA) reimbursement rules (NOTA 1 and 48).

ELIGIBILITY:
All the GPs in Caserta and Bergamo will be invited to participate to the study by the local authorities.

Inclusion Criteria for GPs patients:

* user of Proton Pump Inhibitors (at least one prescriptions in the period of interest)
* aged 65 or above

Exclusion Criteria:

- nursing homes residents

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 800 (Actual)
Dates: Start 2019-10-10 (Actual); Primary Completion 2023-03-14 (Actual); Study Completion 2024-03-14 (Actual)

PRIMARY OUTCOMES:
Short-term effectiveness | 6 months
  Evaluate the short-term (6 months) effectiveness of a low-cost informative intervention in order to improve the appropriateness of prescription of PPI in older people in primary care in agreement with AIFA reimbursement rules by NHS in comparison to the daily clinical practice. Generalised linear mixed model, with a proper link function, on the differences in the proportion of inappropriate prescriptions of PPIs after 6 months from intervention with respect to the baseline, will be used to assess the intervention effectiveness.

SECONDARY OUTCOMES:
Long-term effectiveness | 12-18 months
  Evaluation of the persistence of the effectiveness of the intervention in the long-term at 12 and 18 months. Generalised linear mixed model, with a proper link function, on the differences in the proportion of inappropriate prescriptions of PPIs after 12-18 months from intervention with respect to the baseline, will be used to assess the intervention effectiveness.

OTHER OUTCOMES:
Rate of 'paradoxical effect' | 12-18 months
  Evaluate the rate of 'paradoxical effect' (rebound acid hyper secretion) after gradual cessation of PPI therapy and the rate of the most frequent AEs (i.e. pneumonia, bone fractures, bacterial enteric infections, diminished vitamin absorption, gastric and colon cancer, myocardial infarction and overall mortality ).

CONTACTS AND LOCATIONS:
Overall Officials: Carlotta Franchi, PhD, Principal Investigator — Mario Negri Institute for Pharmacological Research
Locations (3):
- Italy (3):
  - IRCCS MultiMedica- MultiMedica Spa, Sesto San Giovanni, Milan
  - Mario Negri Institute for Pharmacological Research, Milan
  - Università degli studi di Napoli Federico II, Napoli